CLINICAL TRIAL: NCT00504335
Title: A Dose Escalation Trial Evaluating the Safety and Pharmacokinetic Profiles of BIO 300 Capsules in Healthy Male and Female Volunteers
Brief Title: Safety and Pharmacokinetic Study of BIO 300 Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanetics Corporation (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MARC006-025
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Acute Radiation Syndrome
Keywords: Acute Radiation Syndrome; Hematopoietic Syndrome; Radiation Injury; BIO 300
MeSH Terms: conditions — Acute Radiation Syndrome; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 500 BIO 300 capsule (Experimental): The first cohort will receive one 500 BIO 300 capsule and pharmacokinetic blood sampling will be conducted over the first 4 days in an outpatient setting
  Interventions: Drug: BIO 300 Capsules
- 1000 BIO 300 capsule (Experimental): the second cohort will be treated with 1000 mg BIO 300 using the same PK sampling program
  Interventions: Drug: BIO 300 Capsules
- 1500 BIO 300 capsule (Experimental): the third cohort will be treated with 1500 mg BIO 300using the same PK sampling program
  Interventions: Drug: BIO 300 Capsules
- 2000 BIO 300 capsule (Experimental): the forth cohort will be treated with 2000 mg BIO 300using the same PK sampling program
  Interventions: Drug: BIO 300 Capsules

INTERVENTIONS:
Drug: BIO 300 Capsules

SUMMARY:
This trial is designed to evaluate the safety and pharmacokinetics of BIO 300 capsules when administered orally to healthy male and female volunteers. BIO 300 is expected to be safe for use starting at 500 mg.

DETAILED DESCRIPTION:
This clinical trial will assess the safety and PK of BIO 300 capsules at doses expected to deliver a radioprotective or therapeutic effect in humans. Humanetics is planning to conduct this Phase I, single dose, dose-escalation (500, 1000, 1500, and 2000 milligrams) study of the safety, tolerability and pharmacokinetics of BIO 300 by recruiting approximately 24 healthy men and women between the ages of 18 and 64 to be enrolled in cohorts of 6 subjects per group. The first cohort will receive one 500 mg BIO 300 capsule and pharmacokinetic blood sampling will be conducted over the first 4 days in an outpatient setting at a clinic skilled in this type of Phase I trial. Blood samples will be analyzed for BIO 300 levels, hematology, chemistry, lipid profiles, phosphorus, clotting factors and fibrinogen as well as pancreatic lipase and amylase. Urinalysis will assess kidney function as well as creatinine clearance and BIO 300 clearance. All subjects will be monitored for adverse events and the safety of BIO 300 capsules will be evaluated in this setting. After review of all safety information and provided no clinically significant negative findings are revealed, the second cohort will be treated with 1000mg BIO 300 (two 500mg capsules) using the same PK sampling program. Again safety concerns will be reviewed and provided no clinically significant negative findings are revealed, the third and fourth cohort will be treated with 1500 and 2000 mg, respectively, of BIO 300 using the same PK sampling program.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, age 18-64, who have signed the consent form

  * Subjects with a body mass index (BMI) 18-30 kg/m2
  * Subjects who are willing to abstain from sex or use a barrier method of birth control (Women 1 week, Men 4 months after leaving the trial)
  * Subjects with a negative pregnancy test and drug screen
  * Subjects with laboratory values within normal limits (CBC/differential, CMP, enzymes, ECG, vital signs, urinalysis)
  * Subjects with ability to comprehend and complete the questionnaires and forms
  * Subjects who are likely to comply with study procedures and test article consumption
  * Subjects whose schedules permit a 10-12 hour stay in the clinic followed by daily evaluations for one week (7 days)
  * Subjects who are available for a 14-day follow up phone call (women) and 4-month follow up phone call (men).
  * Subjects who are likely to abstain from taking unauthorized medications or supplements or participating in any other clinical trial or experimental treatment during this trial
  * Subjects who are likely to follow the low isoflavone diet program

Exclusion Criteria:

* · Subjects with any allergic reaction or sensitivity to soy, isoflavones, or any component of the test article product

  * Subjects who consume >5 alcoholic beverages per week
  * Subjects who are pregnant, lactating, or at risk of becoming pregnant
  * Subjects who have blood (or urine) levels outside the normal range for any of the hepatic, renal, hematologic, lipid or coagulation parameters measured.
  * Subjects on Hormone Replacement Therapy or Birth Control Pills within the past three months.
  * Subjects on any other clinical trial or experimental treatment in the past 3 months
  * Subjects with a history of diabetes (Type 1 or Type 2 diabetes mellitus) or other endocrine disorders, uncontrolled hypertension, prior cerebrovascular accident or seizure disorder, cardiovascular, hepatic or renal disease, active cancer, hematologic disorder, thromboembolic disease, or HIV infection.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by lab work and adverse event monitoring | 1 month for females & 4 months for males

SECONDARY OUTCOMES:
Pharmacokinetic assessment by analyzing patient serum for free and total BIO 300 content at multiple time points. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: John L Zenk, MD, Principal Investigator — Humanetics Corporation